CLINICAL TRIAL: NCT04719273
Title: A Phase II Clinical Trial Evaluating the Combination of Onapristone With Anastrozole for Women With Refractory Hormone Receptor Positive Endometrial Cancer
Brief Title: Onapristone and Anastrozole for the Treatment of Refractory Hormone Receptor Positive Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20P.829
Record Dates: First submitted 2021-01-04; First posted 2021-01-22 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Refractory Endometrial Adenocarcinoma; Refractory Endometrial Carcinoma; Refractory Endometrial Clear Cell Adenocarcinoma; Refractory Endometrial Endometrioid Adenocarcinoma; Refractory Endometrial Mixed Cell Adenocarcinoma; Refractory Endometrial Serous Adenocarcinoma; Refractory Endometrial Undifferentiated Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (onapristone, anastrozole) (Experimental): Patients receive onapristone PO BID and anastrozole PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles (24 months) until November 30, 2023 or in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Extended-release Onapristone; Drug: Anastrozole; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Diagnostic Test: Estrogen Receptor Positive (Positive Estrogen Receptor; ESR Positive; ESR1 Positive; ER Positive; Estrogen Receptor Alpha Positive); Diagnostic Test: Progesterone Receptor Positive ( PGR Positive; PR Positive)

INTERVENTIONS:
Drug: Extended-release Onapristone — Given PO
  Other Names: ER Onapristone
Drug: Anastrozole — Given PO
  Other Names: 120511-73-1, 2,2'-[5-(1H-1,2,4-Triazol-1-ylmethyl)-1,3-phenylene]di(2-methylpropionitrile), Alpha,alpha,alpha', alpha'-tetramethyl-5-(1H-1,2,4-triazol-1-ylmethyl)-1,3-benzenediacetonitrile,; Anastrazole, Anastrozole, Anastrozole, ANASTROZOLE, anastrozole, Arimidex, ICI D1033, ICI-D1033, ZD-1033
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Diagnostic Test: Estrogen Receptor Positive (Positive Estrogen Receptor; ESR Positive; ESR1 Positive; ER Positive; Estrogen Receptor Alpha Positive) — Immunohistochemistry (IHC):Integral : Tissue
  Other Names: Level/Quantity, Other: Greater than or equal to 1 percent
Diagnostic Test: Progesterone Receptor Positive ( PGR Positive; PR Positive) — Immunohistochemistry (IHC)
  Other Names: Level/Quantity, Other: Greater than or equal to 1 percent

SUMMARY:
This phase II trial studies the effect of onapristone and anastrozole in treating patients with hormone receptor positive endometrial cancer that has not responded to previous treatment (refractory). Progesterone and estrogen are hormones that can cause the growth of endometrial cancer cells. Onapristone blocks the use of progesterone by the tumor cells. Anastrozole is a drug that blocks the production of estrogen in the body. Giving onapristone with anastrozole may work better than anastrozole alone in treating patients with hormone receptor positive endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the activity and safety of a pure progesterone receptor (PR) antagonist, extended-release onapristone (onapristone), with anastrozole to treat women with recurrent metastatic estrogen receptor positive (ER+)/progesterone receptor positive (PR+) endometrial carcinoma.

SECONDARY OBJECTIVES:

I. To estimate the disease control rate (DCR). II. To describe duration of response (DOR). III. To evaluate the safety and tolerability. IV. To evaluate quality of life using the Edmonton Symptom Assessment questionnaire.

EXPLORATORY OBJECTIVES:

I. To characterize the ER and PR expression by immunohistochemistry (IHC) pre- and post-treatment.

OUTLINE:

Patients receive onapristone orally (PO) twice daily (BID) and anastrozole PO once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 24 cycles (24 months) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 1 year after last treatment administration.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Histologically confirmed diagnosis of endometrial cancer with ER and/or PR expression >= 1% by IHC on archival tissue taken within the prior 3 years or new biopsy if no archival tissue is available. IHC results do not have to be from Thomas Jefferson University
* Patients who have failed one prior treatment with a platinum/taxane chemotherapy regimen for management of disease

  * Patients cannot have treatment with more than 2 prior lines of therapy (one line must be platinum/taxane regimen)
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v.)1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension. Each lesion must be >= 10 mm when measured by computed tomography (CT) or magnetic resonance imaging (MRI). Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients with the following histologic epithelial cell types are eligible:

  * Endometrioid adenocarcinoma
  * Serous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Adenocarcinoma not otherwise specified (NOS)
  * Please note: patients with carcinosarcoma are ineligible for this trial
* Patients must have had one prior treatment with a platinum/taxane chemotherapy regimen for management of disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Must have a life expectancy of at least 12 weeks as judged by the treating physician
* Females are only eligible for this study if they are postmenopausal. This is defined as meeting one of the following criteria:

  * S/p total abdominal hysterectomy and bilateral salpingo-oopherectomy
  * Patients who are in menopause is defined clinically as 12 consecutive months of amenorrhea in a woman over 55 in the absence of other biological or physiological causes OR women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Body weight > 30 kg
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl)
* Endocrine and targeted therapy protocols usually enroll patients with aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) in patients without underlying liver metastasis and < 5.0 x ULN in patients with underlying liver metastasis
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or measured creatinine clearance using 24 hours urine collection
* International normalized ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* All subjects must be able to comprehend and sign a written informed consent document
* Resolution of all acute toxic effects of prior therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) grade =< 1, with the exception of unresolved grade 2 neuropathy and grade 2 alopecia, which are allowed
* Patient has recovered from any prior radiotherapy
* Patients must be able to swallow tablets whole, without crushing
* Be able to read and speak English

Exclusion Criteria:

* Concurrent or recent chemotherapy, radiotherapy, immunotherapy, or general anesthesia/major surgery within 3 weeks
* History of prior hormonal therapy (i.e., megestrol acetate, tamoxifen or aromatase inhibitors) for treatment cancer within the past 2 months. Other concurrent hormonal therapy will not be allowed on this trial
* Patient has a concurrent malignancy or history of invasive malignancy within 3 years of enrollment, with the exception of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix that has completed curative therapy
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior systemic anti-cancer therapy including investigational agents within 3 weeks prior to randomization
* Known brain metastasis which have not been treated or showed stability for >= 6 months
* Proteinuria > 1+ on urinalysis or > 1 gm/24 hours (hr)
* Known history of New York Heart Association stage 3 or 4 cardiac disease
* A pleural or pericardial effusion of greater than or equal to grade 3 severity
* Women who are pregnant or nursing
* Has an active infection requiring systemic therapy
* Use of any prescription medication during the prior 28 days of first onapristone dosing that the investigator judges is likely to interfere with onapristone activity; specifically strong inhibitors or inducers, or sensitive substrates of cytochrome P450 CYP3A4
* Patients may not be on a concurrent clinical trial, unless approved by investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year post-treatment
  Defined by the percentage of patients with tumor response (complete response [CR] or partial response [PR]) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Progression-Free Survival (PFS) | At 4 months
  4 month PFS is defined as a binary endpoint, from first dose of onapristone and anastrozole to 4 months of therapy as "confirmed progression-free" or "not progression-free" (including cancer progression or censored subjects). Will use the date of first documented disease progression or recurrence, as assessed by using RECIST 1.1 criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Disease Control Rate | Up to 1 year post-treatment
  Defined as best overall response of CR, PR, or stable disease lasting for >= 24 weeks, per RECIST 1.1.
Time to Response | From randomization to first documented response (CR or PR) in months, assessed up to 1 year post-treatment
Duration of Response | From the first date of documented response to progression or death due to endometrial cancer, assessed up to 1 year post-treatment
Type, frequency and severity of adverse events and laboratory abnormalities | Up to 30 days post-treatment
  Adverse events will be graded for severity according to the Common Terminology Criteria for Adverse Events version 5.0.
Quality of Life and pain score | Up to 1 year post-treatment
  Quality of life and pain scores are defined by the Edmonton Symptom Assessment System using nine subjective patient measures of well-being including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath.

OTHER OUTCOMES:
Estrogen receptor and progesterone receptor expression | Up to 1 year post-treatment
  Assessed by immunohistochemistry and represented as a percentage prior to trial initiation and at progression.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Buchanan, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania